CLINICAL TRIAL: NCT05480683
Title: Addition of Pelvic CT with Agatston Calcium Score for Patients with Peyronie Disease May Change Management Decisions in Patients with Calcified Plaque
Brief Title: Pelvic CT with Agatston Calcium Score for Peyronie Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lauren F. Alexander, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-001770
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peyronie Disease
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Targeted CT of pelvis with specific penile anatomical positioning for Peyronie Disease (Experimental): Subject presenting with Peyronie disease signs or symptoms to Mayo Clinic Florida Department of Urology will undergo a targeted noncontrast CT of the pelvis with specific penile anatomical positioning
  Interventions: Diagnostic Test: CT exam

INTERVENTIONS:
Diagnostic Test: CT exam — Noncontrast CT of the pelvis with specific penile anatomical positioning for coverage and with the protocol optimized for application of Agatston calcium scoring post processing.

SUMMARY:
The purpose of this study is to find out how including a CT exam of the penis can help urologists make treatment decisions for patients with calcified Peyronie's disease.

DETAILED DESCRIPTION:
Peyronie disease (PD) affects up to 10% of men with fibrosing penile plaques causing penile pain and progressing to deformity. Calcified plaque develops in up to 20% of these patients, excluding them from medical therapy with collagenase injection and often requiring more extensive surgery for treatment. PDDU identifies plaque distribution and characteristics while the Doppler exam evaluates for any underlying erectile dysfunction. Calcification can make PDDU difficult to identify the full extent of plaque since the shadow caused by calcification may prevent accurate measurement and over or underestimate the plaque size. In addition, the ultrasound exam is operator dependent and requires injection of an agent to induce erection. Since current clinical practice excludes men with any degree of calcification presumed on physical examination or demonstrated on PDDU from receiving injection therapy they may be triaged to surgical management instead. A prior study found the presence of calcifications at ultrasound had odd ratio 1.75 of patient progressing to surgical management, while fibrosis without calcification did not have increased odds of surgical management. Noncontrast pelvis CT provides three dimensional detail of calcified plaque including parts of the penis that are difficult to image with PDDU, and calcification does not have artifact on CT. By adding non-contrast pelvis CT with Agatston calcium scoring to PDDU and clinical parameters of penile deformity, patients may be better stratified into the appropriate treatment pathway.

ELIGIBILITY:
Inclusion Criteria:

* Peyronie Disease with stable curvature considered for therapeutic intervention
* PDDU obtained at clinic visit
* Able to provide informed consent

Exclusion Criteria:

* Implanted penile prosthesis or implanted urethral sphincter that would prevent adequate CT images
* Acute active Peyronie disease that would not be managed with injection or surgical therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Calcium volume of penile plaques | Baseline
  Peyronie plaques with calcification can be identified with noncontrast CT. The Agatston calcium scoring software is used to mark the calcified plaques to measure the calcium volume (mm3)
Calcium score of penile plaques | Baseline
  Peyronie plaques with calcification can be identified with noncontrast CT. The Agatston calcium scoring software is used to mark the calcified plaques to calculate the Agaston calcium score
Treatment plans adjustment after CT | Within 2 weeks of intervention
  Number of treatment plans to be adjusted after CT results. The treatment options for Peyronie's disease are observation, penile traction therapy, oral medication, medication injection, plaque incision, plaque excision, penile plication with graft, penile plication without graft, penile implant with plaque incision and graft, or penile implant with plication. The study urologist plan will be documented before CT results. After CT results the study urologist will or will not adjust the treatment plan.

SECONDARY OUTCOMES:
Calcified plaque number | Baseline
  Peyronie plaques with calcification can be identified with noncontrast CT and with PDDU. The number of calcified plaques (1, 2, 3 or more than 3) will be counted on CT and PDDU.
Calcified plaque length | Baseline
  Peyronie plaques with calcification can be identified with noncontrast CT and with PDDU. The plaque will be measured in the longest axial and transverse dimensions (mm) on CT and on PDDU.
Calcified plaque continuity | Baseline
  Peyronie plaques with calcification can be identified with noncontrast CT and with PDDU. The plaque will be described as continuous or stippled on CT and PDDU by visual assessment

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Alexander, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials